CLINICAL TRIAL: NCT07179029
Title: Anesthesia Induced Myocardial Injury in Non-cardiac Surgery (AIMY)
Acronym: AIMY
Status: Recruiting | Type: Observational
Sponsor: University Hospital Tuebingen (Other)
Responsible Party: Sponsor
Other Study IDs: AIMY
Record Dates: First submitted 2025-09-10; First posted 2025-09-17 (Actual); Last update posted 2025-09-17 (Actual); Status verified 2025-05

CONDITIONS: Perioperative Myocardial Injury
Keywords: troponin; Perioperative myocardial injury

STUDY DESIGN:
Observational Model: Cohort | Time Perspective: Prospective
Biospecimen Retention: Samples With DNA — Blood
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

GROUPS / COHORTS (1):
- Non-Cardiac Surgery: Non-Cardiac Surgery

SUMMARY:
Myocardial injury during non-cardiac surgery (PMI) affects up to 16% of high-risk patients and represents a significant burden on healthcare systems. An acute myocardial infarction is defined by a dynamic increase in cardiac troponin (cTn) above the 99th percentile and is accompanied by clinical signs of myocardial ischemia. Myocardial injury, on the other hand, is characterized by an increase in cardiac troponin, but without meeting the diagnostic criteria for myocardial infarction. In the perioperative interval, however, it is irrelevant whether a myocardial infarction according to the universal definition or merely an increase in troponin is present, as there is no difference in mortality between the two patient groups. The comprehensive study by Botto et al. provides valuable insights into the severity of MINS and found that 8.0% of patients met the diagnostic criteria. An important finding of this study is that the majority of MINS cases (87.1%) occurred within the first two days after surgery, highlighting the immediate risk of the condition (Botto et al., 2014).

We would like to emphasize the necessity of our prospective, multicenter observational study by highlighting anesthesia-dependent variables such as hemodynamics, type of medication, their potential role, and surgical aspects such as duration of surgery, which represent risk factors for MINS. Identifying and understanding modifiable and non-modifiable risk factors is essential for targeted preoperative intervention. Understanding these factors is crucial for subsequent interventional studies and can also provide criteria for increased monitoring of high-risk patients, as suggested in the current guidelines.

ELIGIBILITY:
Inclusion Criteria:

* Elective or emergency non-cardiac surgery
* Cardiovascular risk: At least two of the following: Age >60 years, hypertension, diabetes mellitus, coronary heart disease, peripheral arterial occlusive disease, cerebrovascular disease, chronic renal insufficiency, chronic heart failure, chronic obstructive pulmonary disease, active smoking
* Age criteria: Adults aged 40-80 years.
* ASA status: ASA classification II-IV.
* Written consent after prior explanation

Exclusion Criteria:

* o Patients unable to give consent: intubated and sedated patients

  * Types of surgery: cardiac surgery, including coronary artery bypass grafting, heart valve repair or replacement, and heart transplantation; obstetric procedures, including cesarean section; minor surgical procedures that do not require general or regional anesthesia (e.g., minor dermatological or ophthalmological procedures)
  * Cardiovascular risk: patients without at least two of the following risk factors: age <40 or >80, no history of hypertension, diabetes, coronary artery disease, peripheral arterial disease, cerebrovascular disease, chronic renal failure, chronic heart failure, chronic obstructive pulmonary disease, and non-smoker status
  * Age criteria: Patients under 40 or over 80 years of age
  * ASA status: ASA classification of I.

Ages: 40 Years to 80 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Study Population: Patients undergoing non- cardiac surgery followed by postoperative blood work
Sampling Method: Probability Sample
Enrollment: 3000 (Estimated)
Dates: Start 2025-05-01 (Actual); Primary Completion 2028-05 (Estimated); Study Completion 2028-05 (Estimated)

PRIMARY OUTCOMES:
Troponin | 1-5 days
  Development of Troponin after non-cardiac surgery
incidence of PMI | 1-5 days
  incidence of PMI after non-cardiac surgery

SECONDARY OUTCOMES:
Mortality | 1-30 days
  Mortality after non-cardiac surgery

CONTACTS AND LOCATIONS:
Overall Officials: Michael Koeppen, MD, Principal Investigator — University Clinic of Tuebingen
Locations (1):
- University Clinic of Tuebingen, Tübingen, Germany

IPD SHARING:
Plan to Share IPD: No